CLINICAL TRIAL: NCT03699800
Title: The Effects of a Graphomotor Intervention Program According to a Psychomotor Approach on Quality and Speed of Handwriting in School-Age Children: A Randomized Controlled Trial
Brief Title: Graphomotor Intervention Program for Handwriting Difficulties Prevention in School-Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Helena Isabel Falcão Coradinho, Principal investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06102018
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Typical Development; Risk of Dysgraphia; Dysgraphia
Keywords: Graphomotor intervention program; Second grade children; Prevention and early identification; Process and product of handwriting; Quality and speed of handwriting
MeSH Terms: conditions — Agraphia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graphomotor intervention program (Experimental): The experimental group (EG) intervention comprises a graphomotor intervention program according to a psychomotor approach. The program integrates two group sessions (6-8 children)/week of 30 minutes for 8 weeks (16 sessions).
  Interventions: Other: Graphomotor intervention program
- Control Group (No Intervention): The control group (CG) participants will maintain their normal classroom activities. After the study, control group participants will be offered the opportunity to integrate a similar graphomotor intervention program.

INTERVENTIONS:
Other: Graphomotor intervention program — The graphomotor intervention program aims to promote the development and reinforcement, different skills involved in the learning process of handwriting and has a preventive character. It follows a bodily, playful, multisensory, exploratory (sensory integration) and neuromotor task training approach and focuses on the following intervention domains: segmental awareness, passive relaxation, trunk-limb dissociation, interdigital coordination, attention, planning, spatial organization/orientation and perception.
  Arms: Graphomotor intervention program

SUMMARY:
12-30% of children present handwriting difficulties, which has negative repercussions on their school career. For this reason, it is fundamental to bet on their prevention. The aim of present study is to examine the effects of a graphomotor intervention program on quality and speed of handwriting in second-grade children. This experimental study is a randomized controlled trial. The program will run for 8 weeks (2 sessions/week of 30 minutes), followed by 6 months of follow-up without intervention. Participants will be assessed 1) at baseline, 2) at the end of the program, and 3) after the follow-up. Participants will be randomly allocated to two groups: experimental group (graphomotor intervention program) and control group.

DETAILED DESCRIPTION:
According to estimates (1), 30% to 60% of the school day is spent performing tasks involving handwriting. It is also in this period that the formal learning of handwriting begins (2). However, not all children are able to develop proficient handwriting (3-4).

According to Alhusaini, Melam and Buragadda (5) 12% to 30% of children present difficulties in handwriting, with negative consequences for school success (6).

Children who fail to develop proficient handwriting are entitled to "poor writers" or "dysgraphics" (7-8).

Dysgraphia refers to a "disturbance or difficulty in the production of written language related to the mechanics of writing" (9). Ajuriaguerra (8) defines it as a writing whose quality is deficient, without any neurological or intellectual deficit explaining it. Generally, handwriting is less legible and organized, contains more erasures and corrections, and exhibits a slower speed (9).

In addition, this is one of the main reasons for referral and consultation in psychomotricity in school-age (10), for this reason it is fundamental to bet on the prevention of them.

The need for prevention and early intervention is indisputable (11). Several studies indicate that both the benefits of late intervention are well-known, because the time is often difficult to correct handwriting difficulties (12-13).

Most of the existing studies focus on remediation of handwriting (14). There is evidence of its efficacy in handwriting improvement, depending on its duration, frequency and method of treatment (5, 7, 15).

There are few studies dedicated to the prevention of handwriting difficulties (14). In addition, to my knowledge, there is no study whose intervention is based on a psychomotor approach. Based on this, a graphomotor intervention program with a psychomotor approach was developed, by Matias and Vieira (16), who will apply in this study to children in the second grade of elementary school.

ELIGIBILITY:
Inclusion Criteria:

* Children in the second grade (aged 7 years old);
* Participation agreement;

Exclusion Criteria:

* Diagnosed or suspected of neurological disabilities (e.g., cerebral palsy, epilepsy), psychiatric and/or behavioural disorders;
* Presence of uncorrected vision and hearing problems;
* Referenced by Special Education/National Service of Early Intervention in Childhood;
* Presence of one or more school retentions;
* Native language is not Portuguese;
* Children with direct intervention in graphomotor skills or who had a similar intervention to that proposed less than 1 year ago;
* Participation in the intervention program of less than 80%;
* Children undergoing drug therapy (e.g., antihistamines) that interfere with the study variables;
* Do not wish to participate in the study.

Ages: 7 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline, between and within groups comparison, in Motor Performance | 0, 4, 10 months
  Outcome Measure - Movement Assessment Battery for Children - Second Edition to assess manual dexterity, aiming and catching and balance
Change from Baseline, between and within groups comparison, in handwriting performance | 0, 4, 10 months
  Outcome Measure - The Concise Assessment Scale for Children's Handwriting (BHK) to assess quality and speed of handwriting
Change from Baseline, between and within groups comparison, in Computerized Handwriting Process Measures | 0, 4, 10 months
  Outcome Measure - The MovAlyzeR to assess spatial, temporal and kinematic variables of handwriting

SECONDARY OUTCOMES:
Sociodemographic characteristics | 0 months
  The Sociodemographic Questionnaire collects data on the identification of the child, the parents, the sociodemographic context and the socioeconomic status of the family based on the Graffar Social Classification Scale Adapted
Change from Baseline, between and within groups comparison, in Manual Preference | 0, 4, 10 months
  Outcome Measure - Manual Preference Questionnaire to assess manual preference

CONTACTS AND LOCATIONS:
Overall Officials: Helena IF Coradinho, MSc, Principal Investigator
Locations (1):
- Helena Isabel Falcão Coradinho, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engel-Yeger B, Rosenblum S. The effects of protracted graphomotor tasks on tripod pinch strength and handwriting performance in children with dysgraphia. Disabil Rehabil. 2010;32(21):1749-57. doi: 10.3109/09638281003734375. PMID 20373859
- [Background] Zeziger P, Deonna T, Mayor C. L'acquisition de l'écriture. Enfance. 2000; 3:295-304. Available at: http://www.persee.fr/doc/enfan_0013-7545_2000_num_53_3_3186
- [Background] Denton PL, Cope S, Moser C. The effects of sensorimotor-based intervention versus therapeutic practice on improving handwriting performance in 6- to 11-year-old children. Am J Occup Ther. 2006 Jan-Feb;60(1):16-27. doi: 10.5014/ajot.60.1.16. PMID 16541981
- [Background] Schneck C, Amundson S. Prewriting and Handwriting Skills. In Case-Smith J., O'Brien J, cords. Occupational Therapy for Children. Missouri: Elsevier; 2010. p. 555-82.
- [Background] Alhusaini AA, Melam GR, Buragadda S. Short-term sensorimotor-based intervention for handwriting performance in elementary school children. Pediatr Int. 2016 Nov;58(11):1118-1123. doi: 10.1111/ped.13004. Epub 2016 Jul 7. PMID 27085075
- [Background] Soppelsa R, Albaret JM. Caractéristiques de la dysgraphie ou du trouble de l'apprentissage de la graphomotricité (TAG) au collège. A.N.A.E. 2014 Fev; 128:1-6. Available at: http://www.psychomot.ups-tlse.fr/Soppelsa-Albaret2014.pdf
- [Background] Rosenblum S, Aloni T, Josman N. Relationships between handwriting performance and organizational abilities among children with and without dysgraphia: a preliminary study. Res Dev Disabil. 2010 Mar-Apr;31(2):502-9. doi: 10.1016/j.ridd.2009.10.016. Epub 2009 Nov 27. PMID 19945252
- [Background] Soppelsa R, Abizeid C, Chéron A, Laurent A, Danna J, Albaret, JM. Dysgraphies et rééducation psychomotrice: Données actuelles. In: Albaret JM, Matta Abizeid C, Soppelsa R. Les Entretiens de Bichat. Publisher: Toulouse - Europa Digital & Publishing, Editors; 2016. p 5-11.
- [Background] Rosenblum S, Dror G. Identifying Developmental Dysgraphia Characteristics Utilizing Handwriting Classification Methods. IEEE Transactions on Human-Machine Systems. 2016 Oct; 47(2): 293-8. doi: 10.1109/THMS.2016.2628799
- [Background] Lachaux-Parker C. Troubles de l'écriture et psychomotricité. Revue francophone d'orthoptie. 2012; 5:143-7. doi: 10.1016/j.rfo.2013.02.002
- [Background] Borghese NA, Palmiotto C, Essenziale J, Mainetti R, Granocchio E, Molteni B et al. Assessment of Exergames as Treatment and Prevention of Dysgraphia. In: Ibáñez J, González-Vargas J, Azorín J, Akay M, Pons J. Converging Clinical and Engineering Research on Neurorehabilitation II. Cham: Springer; 2017. p. 431-6.
- [Background] Graham S, Harris KR. Preventing Writing Difficulties: Providing Additional Handwriting and Spelling Instruction to At-Risk Children in First Grade. Teaching Exceptional Children. 2006 May/Jun; 38(5):64-66. doi: 10.1177/004005990603800509
- [Background] Graham S, Harris KR, & Fink B. Is handwriting causally related to learning to write? Treatment of handwriting problems in beginning writers. Journal of Educational Psychology. 2000; 92(4):620-33. doi: 10.1037/0022-0663.92.4.620
- [Background] Howe TH, Roston KL, Sheu CF, Hinojosa J. Assessing handwriting intervention effectiveness in elementary school students: a two-group controlled study. Am J Occup Ther. 2013 Jan-Feb;67(1):19-26. doi: 10.5014/ajot.2013.005470. PMID 23245779
- [Background] Hoy MM, Egan MY, Feder KP. A systematic review of interventions to improve handwriting. Can J Occup Ther. 2011 Feb;78(1):13-25. doi: 10.2182/cjot.2011.78.1.3. PMID 21395194
- [Background] Matias A, Vieira C. Programa de intervenção grafomotora. [In press].